CLINICAL TRIAL: NCT04167514
Title: A Randomized, Double-Blind, Placebo-Controlled Multicenter Phase III Trial of Alpha 1 - Antitrypsin (AAT) Combined With Corticosteroids vs Corticosteroids Alone for the Treatment of High Risk Acute Graft-versus-Host Disease (GVHD) Following Allogeneic Hematopoietic Stem Cell Transplant
Brief Title: Treatment of GVHD in Hematopoietic Stem Cell Transplant (HSCT) Recipients Using AAT Plus Corticosteroids (CS) Compared With Corticosteroids Alone
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: CSL Behring (Industry)
Collaborators: Blood and Marrow Transplant Clinical Trials Network (Network); National Institutes of Health (NIH) (NIH); National Heart, Lung, and Blood Institute (NHLBI) (NIH); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CSL964_5001 / BMT CTN 1705; BMT CTN Protocol 1705 (Other: Blood and Marrow Transplant Clinical Trials Network (BMT CTN))
Record Dates: First submitted 2019-11-15; First posted 2019-11-19 (Actual); Results first posted 2025-08-29 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Graft Versus Host Disease (GVHD)
MeSH Terms: conditions — Graft vs Host Disease | interventions — alpha 1-Antitrypsin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- AAT (Experimental): Alpha-1 antitrypsin (AAT) is a lyophilized powder for intravenous administration
  Interventions: Biological: Alpha-1 antitrypsin (AAT)
- Placebo (Placebo Comparator): Albumin solution administered intravenously
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: Alpha-1 antitrypsin (AAT) — AAT is a lyophilized product for intravenous administration
  Other Names: Alpha-1 proteinase inhibitor (A1-P1)
  Arms: AAT
Drug: Placebo — Albumin solution administered intravenously
  Arms: Placebo

SUMMARY:
Study CSL964_5001 will investigate the efficacy of AAT with corticosteroids compared with corticosteroids alone as first line therapy for patients with high-risk acute GVHD

ELIGIBILITY:
Inclusion Criteria:

* Patients 12 years of age or older
* Initial presentation of acute GVHD after allogeneic hematopoietic cell transplantation for any indication
* Any graft or donor source or conditioning intensity
* Clinical diagnosis of acute GVHD requiring systemic therapy with corticosteroids

Exclusion Criteria:

* Prior exogenous AAT exposure for GVHD prophylaxis
* Relapsed, progressing, or persistent malignancy
* de novo chronic GVHD or overlap syndrome developing before or present at the time of enrollment
* Receiving other drugs for the treatment of GVHD
* Receiving systemic CS for any indication within 7 days before the onset of acute GVHD

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 136 (Actual)
Dates: Start 2020-01-09 (Actual); Primary Completion 2023-09-11 (Actual); Study Completion 2024-06-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — CSL Behring
Locations (25):
- United States (25):
  - Stanford University, Stanford, California
  - University of Florida, Gainesville, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Emory University, Atlanta, Georgia
  - Northside Hospital, Atlanta, Georgia
  - IU Hospital, Indianapolis, Indiana
  - Univ. of Kansas Cancer Center, Westwood, Kansas
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - U-M Medical Center, Ann Arbor, Michigan
  - Karmanos Cancer Center, Detroit, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - Washington University, St Louis, Missouri
  - MSKCC, New York, New York
  - Levine Cancer Center, Charlotte, North Carolina
  - Duke, Durham, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - Ohio State Univ.Medical Center, Columbus, Ohio
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - Center for Gene Therapy, Houston, Texas
  - MD Anderson Cancer Center, Houston, Texas
  - Virginia Commonwealth Univ., Richmond, Virginia
  - Fred Hutchinson Clinic, Seattle, Washington
  - University of Wisconsin, Madison, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
CSL will consider on a case-by-case basis requests to share Individual Patient Data (IPD) with external bona-fide, qualified scientific and medical researchers. For information on the process and requirements for submitting a voluntary data sharing request for IPD, please contact CSL at clinicaltrials@cslbehring.com.
Supporting Information: Study Protocol, SAP
Time Frame: Requests for IPD will generally be considered once review by major regulatory authorities (ie FDA, EMA) is complete and the primary publication is available.
Access Criteria: Proposed research should seek to answer a previously unanswered important medical or scientific question.
  Applicable country specific privacy and other laws and regulations will be considered and may prevent sharing of IPD.
  If the request is approved and the researcher has executed an appropriate data sharing agreement, IPD that has been appropriately anonymized will be available.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 26 investigative sites in the United States of America.
Pre-assignment Details: A total of 136 participants were randomized in this study.
Groups:
- Alpha-1 Antitrypsin (AAT): Participants received AAT twice weekly through Day 28. Responding participants (Complete Response/Partial Response [CR/PR]) continued to receive a once weekly dose of AAT through Day 56.
- Placebo: Participants received albumin solution administered intravenously (IV) to match the investigational medicinal product (IMP) twice weekly through Day 28. Responding participants (CR/PR) continued to receive a once weekly dose of matching placebo through Day 56.
Period: Overall Study
Arm/Group | Alpha-1 Antitrypsin (AAT) | Placebo
Started | 65 | 71
Treated | 63 | 69
Completed | 38 | 41
Not Completed | 27 | 30
Not completed — Adverse event, not serious | 0 | 1
Not completed — Lost to Follow-up | 1 | 0
Not completed — Participant Decision | 2 | 4
Not completed — Physician Decision | 3 | 2
Not completed — Death | 14 | 18
Not completed — Enrolled but treatment not administered | 2 | 0
Not completed — Multiple reasons for study discontinuation documented; including death, primary reason not reported | 3 | 1
Not completed — Multiple reasons for study discontinuation documented; excluding death, primary reason not reported | 2 | 4

BASELINE CHARACTERISTICS:
Population: Analysis was performed on the intent-to-treat (ITT) population. The ITT population consisted of all randomized participants, classified according to their randomized treatment assignments. All randomized participants were included, regardless of whether the assigned study treatment was truly administered.
Groups:
- Alpha-1 Antitrypsin (AAT): Participants received AAT twice weekly through Day 28. Responding participants (CR/PR) continued to receive a once weekly dose of AAT through Day 56.
- Placebo: Participants received albumin solution administered IV to match the IMP twice weekly through Day 28. Responding participants (CR/PR) continued to receive a once-weekly dose of matching placebo through Day 56.
- Total: Total of all reporting groups
Arm/Group | Alpha-1 Antitrypsin (AAT) | Placebo | Total
Number analyzed (Participants) | 65 | 71 | 136
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.6 (12.65) | 55.3 (13.75) | 55.9 (13.20)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 32 | 52
  Male | 45 | 39 | 84
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 3 | 11
  Not Hispanic or Latino | 56 | 66 | 122
  Unknown or Not Reported | 1 | 2 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 5 | 2 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 6 | 9
  White | 51 | 61 | 112
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 6 | 2 | 8

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (ORR) to Acute Graft-versus-Host Disease (GVHD) Treatment
Description: The overall response is defined as having a CR or PR at Day 28, along with: being alive, free of any next-line GVHD therapy, and free of escalation of prednisone-equivalent steroid dose to 2.5 milligrams per kilogram (mg/kg)/day or more. The percentage of participants with CR or PR is reported here. Wilson score confidence intervals (CIs) are reported here as a measure of dispersion.
  The CR was defined as a score of 0 for the GVHD staging in all evaluable organs. The PR was defined as an improvement in one or more organs involved with GVHD symptoms without progression in others. Acute GVHD was graded and assessed for response based on Harris (Mount Sinai Acute GVHD International Consortium [MAGIC]) criteria (stage 0, 1, 2, 3, 4) for skin, liver, upper gastrointestinal (GI) tract, and lower GI tract. Participants who had an escalation of prednisone-equivalent steroid dose to 2.5 mg/kg/day or higher were classified as non-responders (NR).
Time Frame: At Day 28
Population: Analysis was performed on the ITT population. The ITT population consisted of all randomized participants, classified according to their randomized treatment assignments. All randomized participants were included, regardless of whether the assigned study treatment was truly administered.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Alpha-1 Antitrypsin (AAT) | Placebo
Number analyzed (Participants) | 65 | 71
percentage of participants | 60.0 [47.86 to 71.03] | 45.1 [34.05 to 56.60]
Statistical Analysis 1: Comparison: Alpha-1 Antitrypsin (AAT) vs Placebo; Test type: Superiority; p = 0.034, One-sided Wald; One-sided Wald test of superior odds of overall response under AAT treatment compared to placebo.Threshold of significance at <0.025; Odds Ratio (OR) = 1.92, 95% CI 2-sided [0.954 to 3.866] — Wald CIs

2. Secondary Outcome: Duration of Response (DOR)
Description: The DOR was defined as time from the Day 28 response (CR or PR) until the first of the following events occurs: progression of acute GVHD, death, any next-line GVHD therapy, or escalation of prednisone-equivalent steroids to greater than or equal to (>=) 2.5 mg/kg/day. Wald CIs are reported here as a measure of dispersion.
Time Frame: Up to 12 months
Population: Analysis was performed on the ITT population participants with a response as defined in the measure description of the primary outcome measure. The ITT population consisted of all randomized participants, classified according to their randomized treatment assignments. All randomized participants were included, regardless of whether the assigned study treatment was truly administered.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Alpha-1 Antitrypsin (AAT) | Placebo
Number analyzed (Participants) | 39 | 32
days | 82 [22 to 176] | 154 [57 to NA] — The upper limit of 95% Confidence interval was not estimable due to low number of events.

3. Secondary Outcome: Number of Participants With Non-relapse Mortality (NRM) Event
Description: An event of NRM was death without prior evidence of relapse/progression of the primary disease, where relapse/progression was treated as a competing risk. Cumulative incidence of NRM at 6 and 12 months post-randomization is reported here for this outcome measure.
Time Frame: At 6 and 12 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Alpha-1 Antitrypsin (AAT) | Placebo
Number analyzed (Participants) | 65 | 71
Participants
  At 6 months | 12 | 14
  At 12 months | 13 | 14

4. Secondary Outcome: Number of Overall and Progression-free Survival Events
Description: An event for overall survival (OS) was death from any cause, while an event for progression-free survival (PFS) was death from any cause or relapse/progression of the primary disease.
Time Frame: At 6 and 12 months
Population: as for outcome 1
Measure: Number; unit: events
Arm/Group | Alpha-1 Antitrypsin (AAT) | Placebo
Number analyzed (Participants) | 65 | 71
events
  OS: At 6 months | 16 | 18
  OS: At 12 months | 20 | 23
  PFS: At 6 months | 25 | 28
  PFS: At 12 months | 27 | 29

5. Secondary Outcome: Number of Participants With GVHD-free Survival
Description: GVHD-free survival was defined as participants being alive, free of acute or chronic GVHD, and free of any next-line GVHD therapy or escalation of steroids to >=2.5 mg/kg/day prednisone or equivalent for treatment of GVHD.
Time Frame: At Day 56
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Alpha-1 Antitrypsin (AAT) | Placebo
Number analyzed (Participants) | 65 | 71
Participants | 29 | 25

6. Secondary Outcome: Percentage of Participants With Response
Description: The percentage of participants with CR, PR (including subset with very good partial response [VGPR]), and treatment failure (TF). The designation of TF consisted of participants with NR, mixed response (MR) or progression. The initiation of additional systemic (next-line) GVHD therapies, escalation of prednisone equivalent steroid dose to >= 2.5 mg/kg/day, or death from any cause prior to the assessment timepoint was also considered a TF. Simultaneous Goodman CIs are provided for category proportions for each arm at each assessment time.
Time Frame: At Day 7, 14, 21, 28, 56, and 86
Population: Analysis was performed on the ITT population. The ITT population consisted of all randomized participants, classified according to their randomized treatment assignments. All randomized participants were included, regardless of whether the assigned study treatment was truly administered. Here, the 'number analyzed' for Day 86 includes responses for only those participants who remained on maintenance treatment after Day 28.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Alpha-1 Antitrypsin (AAT) | Placebo
Number analyzed (Participants) | 65 | 71
percentage of participants
  At Day 7 - CR | 29.2 [17.86 to 43.97] | 33.8 [22.03 to 48.00]
  At Day 7 - PR | 33.8 [21.62 to 48.69] | 25.4 [15.16 to 39.22]
  At Day 7 - TF | 36.9 [24.20 to 51.76] | 40.8 [28.08 to 54.98]
  At Day 14 - CR | 47.7 [33.66 to 62.10] | 46.5 [33.11 to 60.38]
  At Day 14 - PR | 23.1 [13.07 to 37.45] | 14.1 [6.89 to 26.65]
  At Day 14 - TF | 29.2 [17.86 to 43.97] | 39.4 [26.85 to 53.61]
  At Day 21 - CR | 55.4 [40.79 to 69.10] | 40.8 [28.08 to 54.98]
  At Day 21 - PR | 9.2 [3.66 to 21.41] | 9.9 [4.18 to 21.54]
  At Day 21 - TF | 35.4 [22.91 to 50.23] | 49.3 [35.68 to 63.01]
  At Day 28 - CR | 55.4 [40.79 to 69.10] | 40.8 [28.08 to 54.98]
  At Day 28 - PR | 4.6 [1.28 to 15.31] | 4.2 [1.17 to 14.12]
  At Day 28 - TF | 40.0 [26.84 to 54.78] | 54.9 [40.96 to 68.16]
  At Day 56 - CR | 44.6 [30.90 to 59.21] | 35.2 [23.22 to 49.42]
  At Day 56 - PR | 6.2 [2.00 to 17.41] | 4.2 [1.17 to 14.12]
  At Day 56 - TF | 49.2 [35.06 to 63.52] | 60.6 [46.39 to 73.15]
  At Day 86 - CR: number analyzed (Participants) | 41 | 40
  At Day 86 - CR | 63.4 [44.82 to 78.72] | 50.0 [32.30 to 67.70]
  At Day 86 - PR: number analyzed (Participants) | 41 | 40
  At Day 86 - PR | 2.4 [0.32 to 16.22] | 10.0 [3.27 to 26.76]
  At Day 86 - TF: number analyzed (Participants) | 41 | 40
  At Day 86 - TF | 34.1 [19.37 to 52.81] | 40.0 [23.87 to 58.64]

7. Secondary Outcome: Percentage of Participants With Response Allowing for Approved Next-line Therapy
Description: The percentage of participants with CR, PR (including subset with VGPR), and TF allowing for treatment with next-line therapy. The designation of TF consisted of participants with NR, MR, or progression. The escalation of prednisone-equivalent steroid dose to >= 2.5 mg/kg/day or death from any cause prior to the assessment timepoint was also considered a TF. Simultaneous Goodman CIs are provided for category proportions for each arm at each assessment time.
Time Frame: At Day 7, 14, 21, 28, 56, and 86
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Alpha-1 Antitrypsin (AAT) | Placebo
Number analyzed (Participants) | 65 | 71
percentage of participants
  At Day 7 - CR | 29.2 [17.86 to 43.97] | 33.8 [22.03 to 48.00]
  At Day 7 - PR | 36.9 [24.20 to 51.76] | 31.0 [19.69 to 45.12]
  At Day 7 - TF | 33.8 [21.62 to 48.69] | 35.2 [23.22 to 49.42]
  At Day 14 - CR | 50.8 [36.48 to 64.94] | 46.5 [33.11 to 60.38]
  At Day 14 - PR | 29.2 [17.86 to 43.97] | 26.8 [16.27 to 40.72]
  At Day 14 - TF | 20.0 [10.79 to 34.07] | 26.8 [16.27 to 40.72]
  At Day 21 - CR | 56.9 [42.26 to 70.47] | 46.5 [33.11 to 60.38]
  At Day 21 - PR | 15.4 [7.54 to 28.84] | 18.3 [9.85 to 31.51]
  At Day 21 - TF | 27.7 [16.63 to 42.37] | 35.2 [23.22 to 49.42]
  At Day 28 - CR | 63.1 [48.24 to 75.80] | 49.3 [35.68 to 63.01]
  At Day 28 - PR | 9.2 [3.66 to 21.41] | 14.1 [6.89 to 26.65]
  At Day 28 - TF | 27.7 [16.63 to 42.37] | 36.6 [24.41 to 50.82]
  At Day 56 - CR | 52.3 [37.90 to 66.34] | 47.9 [34.39 to 61.70]
  At Day 56 - PR | 13.8 [6.52 to 27.03] | 4.2 [1.17 to 14.12]
  At Day 56 - TF | 33.8 [21.62 to 48.69] | 47.9 [34.39 to 61.70]
  At Day 86 - CR: number analyzed (Participants) | 41 | 40
  At Day 86 - CR | 65.9 [47.19 to 80.63] | 72.5 [53.62 to 85.74]
  At Day 86 - PR: number analyzed (Participants) | 41 | 40
  At Day 86 - PR | 7.3 [2.04 to 23.07] | 10.0 [3.27 to 26.76]
  At Day 86 - TF: number analyzed (Participants) | 41 | 40
  At Day 86 - TF | 26.8 [13.90 to 45.45] | 17.5 [7.52 to 35.63]

8. Secondary Outcome: Incidence of Grade 2 to 3 Systemic Infections
Description: The cumulative incidence of Grade 2 to 3 systemic infections. Grade 2 to 3 systemic infections were defined according to the Blood and Marrow Transplant Clinical Trials Network (BMT CTN) Manual of Procedures.
Time Frame: Up to 90 days (including 30 days after last dose of study drug)
Population: Analysis was performed on the safety population. The safety population included all randomized participants who received at least one dose of study treatment. Participants were classified according to the treatment received.
Measure: Number; unit: events
Arm/Group | Alpha-1 Antitrypsin (AAT) | Placebo
Number analyzed (Participants) | 63 | 69
events | 20 | 22

9. Secondary Outcome: Percentage of Participants With Grade 3 to 5 Treatment-emergent Adverse Events (TEAEs)
Description: The incidence of Grade 3 to 5 TEAEs (per Common Terminology Criteria for Adverse Events [CTCAE] Version 5.0). Wilson score CIs are reported here as a measure of dispersion.
Time Frame: Up to 30 days after the last dose of study drug
Population: as for outcome 8
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Alpha-1 Antitrypsin (AAT) | Placebo
Number analyzed (Participants) | 63 | 69
percentage of participants | 46.0 [34.31 to 58.21] | 65.2 [53.45 to 75.38]

10. Secondary Outcome: Cumulative Incidence of Chronic GVHD
Description: Chronic GVHD was defined per National Institutes of Health (NIH) Consensus Criteria. Diagnosis of chronic GVHD of any severity (mild, moderate, or severe) was considered an event for this outcome measure, where death before cGVHD was treated as a competing risk.
Time Frame: At 6 and 12 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Alpha-1 Antitrypsin (AAT) | Placebo
Number analyzed (Participants) | 65 | 71
Participants
  At 6 months | 13 | 9
  At 12 months | 20 | 14

11. Secondary Outcome: Cumulative Incidence of Disease Relapse/ Progression of Primary Disease
Description: The cumulative incidence of relapse/progression of the primary disease, with death prior to relapse/progression treated as a competing risk. Death without prior relapse/progression was treated as a competing risk for relapse/progression.
Time Frame: At 6 months and 12 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Alpha-1 Antitrypsin (AAT) | Placebo
Number analyzed (Participants) | 65 | 71
Participants
  At 6 months | 14 | 14
  At 12 months | 15 | 15

12. Other Pre Specified Outcome: DOR - Supplementary Analysis
Description: The DOR was defined as time from the Day 28 response (CR or PR) until the first of the following events occurs: death, any next-line GVHD therapy, or escalation of prednisone-equivalent steroids to >= 2.5 mg/kg/day. Wald CIs are reported here as a measure of dispersion.
Time Frame: Up to 12 months
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Alpha-1 Antitrypsin (AAT) | Placebo
Number analyzed (Participants) | 39 | 32
days | NA [85 to NA] — The median and upper limit of 95% CI were not estimable due to low number of events. | NA [109 to NA] — The median and upper limit of 95% CI were not estimable due to low number of events.

ADVERSE EVENTS:
Time Frame: From randomization to 12 months (end of study [EOS] follow-up): AEs and Serious AEs (SAEs) reported from randomization until 30 days post last dose. Beginning at 31 days from the last dose of the study drug through the EOS follow-up, only SAEs related to the study drug and unanticipated SAEs (regardless of relationship) required reporting. All-cause mortality includes any deaths, regardless of the timing, including those reported beyond the 12 months, up to 16 months for the last reported death.
Description: All-cause mortality data are presented for the ITT population, which consisted of all randomized participants, classified according to their randomized treatment assignments. Analysis of serious AEs (SAEs) and non-serious AEs was performed on the safety population, which included all randomized participants who received at least one dose of study treatment.
Arm/Group | Alpha-1 Antitrypsin (AAT) | Placebo
All-Cause Mortality (participants affected / at risk) | 21/65 | 23/71
Serious Adverse Events (participants affected / at risk) | 11/63 | 23/69
Other Adverse Events (participants affected / at risk) | 37/63 | 42/69
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Alpha-1 Antitrypsin (AAT) (N=63) | Placebo (N=69)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 4 (4)
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Vascular access complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Intracranial mass (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Toxic encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1)
Depressed level of consciousness (Nervous system disorders) | 0 (0) | 1 (1)
Encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Metabolic encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Small intestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Failure to thrive (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Thrombotic microangiopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Autoimmune haemolytic anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Haemolytic uraemic syndrome (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Methaemoglobinaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Atrial tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial ischaemia (Cardiac disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (2)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 2 (2) | 0 (0)
Asthenia (General disorders) | 1 (2) | 0 (0)
Multiple organ dysfunction syndrome (General disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
Embolism (Vascular disorders) | 0 (0) | 1 (1)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 1 (1)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatic failure (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hallucination (Psychiatric disorders) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 2 (2)
Transaminases increased (Investigations) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Alpha-1 Antitrypsin (AAT) (N=63) | Placebo (N=69)
Hyperglycaemia (Metabolism and nutrition disorders) | 13 (15) | 11 (15)
Hypomagnesaemia (Metabolism and nutrition disorders) | 10 (15) | 10 (23)
Hypocalcaemia (Metabolism and nutrition disorders) | 7 (16) | 12 (26)
Hyperkalaemia (Metabolism and nutrition disorders) | 6 (11) | 9 (13)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 9 (27) | 6 (12)
Hyponatraemia (Metabolism and nutrition disorders) | 6 (12) | 9 (16)
Hypophosphataemia (Metabolism and nutrition disorders) | 8 (15) | 5 (10)
Hypokalaemia (Metabolism and nutrition disorders) | 6 (9) | 5 (8)
Decreased appetite (Metabolism and nutrition disorders) | 3 (3) | 6 (6)
Hyperphosphataemia (Metabolism and nutrition disorders) | 3 (3) | 4 (4)
Hypermagnesaemia (Metabolism and nutrition disorders) | 2 (2) | 4 (4)
Alanine aminotransferase increased (Investigations) | 7 (8) | 11 (17)
Aspartate aminotransferase increased (Investigations) | 5 (10) | 8 (12)
Blood alkaline phosphatase increased (Investigations) | 4 (5) | 8 (12)
Blood bilirubin increased (Investigations) | 4 (6) | 6 (8)
Blood creatinine increased (Investigations) | 4 (4) | 6 (8)
Blood lactate dehydrogenase increased (Investigations) | 5 (6) | 5 (9)
Abdominal pain (Gastrointestinal disorders) | 9 (10) | 6 (6)
Dry mouth (Gastrointestinal disorders) | 7 (9) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 4 (4)
Constipation (Gastrointestinal disorders) | 4 (6) | 1 (1)
Oedema peripheral (General disorders) | 12 (13) | 10 (12)
Fatigue (General disorders) | 5 (5) | 7 (9)
Hypertension (Vascular disorders) | 9 (12) | 10 (16)
Hypotension (Vascular disorders) | 6 (9) | 3 (3)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6 (9) | 8 (8)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 4 (4)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (4) | 4 (5)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 5 (5) | 8 (9)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 (5) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 6 (6)
Tremor (Nervous system disorders) | 4 (4) | 2 (2)
Insomnia (Psychiatric disorders) | 4 (4) | 6 (6)
Fall (Injury, poisoning and procedural complications) | 2 (2) | 6 (6)
Anaemia (Blood and lymphatic system disorders) | 5 (20) | 2 (9)
Sinus tachycardia (Cardiac disorders) | 4 (9) | 3 (3)
Dysuria (Renal and urinary disorders) | 4 (4) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2023-09-22): https://cdn.clinicaltrials.gov/large-docs/14/NCT04167514/Prot_000.pdf
  • Statistical Analysis Plan (2024-02-08): https://cdn.clinicaltrials.gov/large-docs/14/NCT04167514/SAP_002.pdf